CLINICAL TRIAL: NCT06097871
Title: A Double-Blinded, Randomized Control Evaluation of the Efficacy of an Oral Acne Supplement for Adult Women
Brief Title: RCT of an Oral Acne Supplement for Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceutical Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NW-CS-03
Record Dates: First submitted 2023-10-16; First posted 2023-10-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: 1-1 randomization to placebo or active treatment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the subject and the investigator will be blinded to the subject's group allocation. All outcomes will be assessed by the blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutraceutical Dietary Supplement (Experimental): A novel nutraceutical skin supplement, scientifically formulated to specifically target the multiple underlying causes of acne in women. The supplement is comprised of primary and secondary ingredients, designed to improve skin from the inside out.
  Interventions: Dietary Supplement: Skin Nutraceutical Supplement
- Placebo (Placebo Comparator): Oral supplement containing non-active ingredients.
  Interventions: Other: Placebo pill

INTERVENTIONS:
Dietary Supplement: Skin Nutraceutical Supplement — The Skin Nutraceutical Supplement is made with Nutrafol's patented Synergen Skin Complex®, which is a blend of proprietary formulation of botanicals with potent anti-inflammatory, anti-stress adaptogenic, antioxidant and DHT-inhibiting properties combined to synergistically combat the multiple underlying factors that compromise skin health. These ingredients include Holy Basil, Maca, Curcumin, and Berberine in combination with other nutrients used to support skin health such as olive extract (20% hydroxytyrosol), konjac root (3% ceramides), vitamin A, B vitamins, and vitamin C.
  Arms: Nutraceutical Dietary Supplement
Other: Placebo pill — A placebo pill containing non-active ingredients
  Arms: Placebo

SUMMARY:
This study is to assess the efficacy and tolerability of an oral supplement in mild to moderate acne in adult females.

DETAILED DESCRIPTION:
This is a 12-week, single-center, placebo controlled double blind, randomized clinical trial in adult female subjects with mild to moderate non-cystic acne. Female subjects will be enrolled in this single site study to evaluate the efficacy of an oral acne supplement. Upon enrollment, subjects will be randomized to a treatment or a placebo group. Both the subject and the investigator will be blinded to the subject's group allocation. The objective of this research is to assess the efficacy and tolerability of an oral supplement in mild to moderate non-cystic acne in adult females when compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Females subjects 18-50 years of age.
2. Subjects with mild to moderate (non-cystic) acne (8 inflammatory lesions, 10 non-inflammatory lesions).
3. Subjects with an IGA score of 2-3
4. Subjects with all skin types (normal, oily, etc.)
5. Subjects with all Fitzpatrick skin types I-VI.
6. Subjects who agree to use only the provided study skin cleansing, moisturizing, and sunscreen products during the study duration.
7. Subjects agree not to introduce any new colored cosmetics (lipsticks, eye shadows, facial foundations, blush, powder) on their face.
8. No known medical conditions that, in the investigator's opinion, may interfere with study participation.
9. Women of childbearing potential must be willing to use a form of birth control during the study. For the purpose of this study, the following are considered acceptable methods of birth control: oral contraceptives, Norplant®, Depo-Provera®, double barrier methods (e.g., condom and spermicide) and abstinence.
10. Subjects are dependable and able to follow directions and willing to comply with the schedule of visits.
11. Subjects in generally good physical and mental health.
12. Able to read, write, speak, and understand English
13. Individual (and/or his/her legally acceptable representative, as applicable) has signed the Consent for Photograph Release and ICD including Health Insurance Portability and Accountability Act (HIPAA) disclosure.
14. Subject must avoid sun exposure.
15. Subject must avoid professional or facial spa procedures during the study.

Exclusion Criteria:

1. Any dermatological disorder, which in the investigator's opinion, may interfere with the accurate evaluation of the subject's skin characteristics, except for the study condition of acne.
2. Subjects who are not willing to use the assigned skin care study products to their face as instructed and are not willing to take an oral acne supplement.
3. Females who are pregnant, lactating, or planning to become pregnant during the study or within 30 days of study completion. (Subject must document her response in either the source documentation or informed consent/assent forms).
4. Subject has a surgery and/or invasive medical procedure planned during the study.
5. Subject has observable suntan, scars, nevi, tattoo, excessive hair (including beard, mustache, or goatee), or other dermal conditions on the face that could interfere with study evaluations or confound study results, as determined by the PI or designee.
6. Subject has a history of or a concurrent health condition/situation which, in the opinion of the PI, if medically qualified, or study physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study.
7. Subject is an employee/contractor or immediate family member of the PI, Study Site, or Sponsor.
8. Subjects with clinically significant unstable medical disorders.
9. Subjects who are unwilling or unable to comply with the requirements of the protocol.
10. Subjects with any known allergies or sensitivities to the study products.
11. Subjects who have a history of a psychological illness or condition that would interfere with their ability to understand and follow the requirements of the study.
12. Subjects who have acne nodules/cysts representative of severe acne.
13. Subjects who are currently using, planning to use during the study or has used any of the following in the specified time range (based on subject report):

    * 1 month prior to Visit 1: Prescription (oral or topically applied on the face) antibiotics, inhaled steroids (except those prescribed for allergies), or hormones (pre- or post-menopausal hormone-replacement therapy; insulin, etc.), or other medications that could make skin more sensitive or have an effect on the skin, as determined by the PI or designee. Oral contraceptives are acceptable.
    * 1 month prior to Visit 1: Prescription medication for acne (e.g. doxycycline, minocycline, clindamycin, sulfamethoxazole and trimethoprim [Bactrim], tetracycline, erythromycin, azithromycin, or Vibramycin®)
    * 1 month prior to Visit 1: Topical prescription retinoids (e.g. Retin-A®, Retin-A Micro®, Renova®, Adapalene, Tazarotene, Avita®, Tazorac®, Avage®, Differin®), azelaic acid, benzoyl peroxide, dapsone, sodium sulfacetamide, Epiduo®, or other similar prescription drug on the face
    * 6 months prior to Visit 1: Accutane or other oral retinoid
    * 2 weeks prior to Visit 1: Any of the following on the face:

      * Light therapy
      * OTC topical medications/products (including antiacne or antibacterial agents, topical anti-inflammatories, topical retinoids, etc.). Sunscreens (SPF) are acceptable.
14. Subject is taking medications that would mask an adverse event (AE) or influence the study results, including:

    * Immunosuppressive drugs and steroidal and/or non-steroidal anti-inflammatory drugs within 3 months before Visit 1 and during the study.
    * Regular use of antihistamines within 1 month before Visit 1 and during the study.
15. Subject has a history of or a concurrent health condition/situation, which in the opinion of the PI, if medically qualified, or Study Physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study.
16. Subjects who are currently experiencing an acne flare.
17. Subjects having started hormone replacement therapies (HRT) or hormones for birth control less than 3 months prior to the study entry or who plan on starting, stopping or changing doses of HRT or hormones for birth control during the study.
18. Subjects taking any medication or supplement that has a known interaction with any of the study product ingredients, including but not limited to Berberine, which is associated with inhibition of CYP450 enzymes.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
Change in IGA at 12 weeks | 12 weeks
  The primary efficacy endpoint is the investigator assessed change from baseline to week 12 in facial acne IGA rating compared to placebo.

SECONDARY OUTCOMES:
Change in IGA at 4 weeks | 4 weeks
  Investigator assessed change from baseline to week 4 in facial acne IGA rating compared to placebo
Change in IGA a 8 weeks | 8 weeks
  Investigator assessed change from baseline to week 8 in facial acne IGA rating compared to placebo
Change in corneometry measurements at 4 weeks | 4 weeks
  Change in corneometry measurements from baseline to week 4 compared to placebo.
Change in sebumeter measurements at 4 weeks | 4 weeks
  Change in sebumeter measurements from baseline to week 4 compared to placebo.
Change in corneometry measurements at 8 weeks | 8 weeks
  Change in corneometry measurements from baseline to week 8 compared to placebo.
Change in sebumeter measurements at 8 weeks | 8 weeks
  Change in sebumeter measurements from baseline to week 8 compared to placebo.
Change in corneometry measurements at 12 week | 12 weeks
  Change in corneometry measurements from baseline to week 12 compared to placebo.
Change in sebumeter measurements at 12 week | 12 weeks
  Change in sebumeter measurements from baseline to week 12 compared to placebo.
Subject assessed improvement at week 4 | 4 weeks
  Subject assessed improvement in using a self assessment questionnaire at week 4 compared to placebo.
Subject assessed improvement at week 8 | 8 weeks
  Subject assessed improvement in using a self assessment questionnaire week 8 compared to placebo.
Subject assessed improvement at week 12 | 12 weeks
  Subject assessed improvement using a self assessment questionnaire at week 12
Product-Related Safety outcomes | All visits until 12 weeks
  Overall incidence of all study product-related adverse events reported during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Draelos Z, Harper J, Farris PK, Hazan A, Raymond I. A 12-Week Randomized, Double-Blind, Placebo-Controlled Trial for the Efficacy and Safety of a Novel Nutraceutical for Mild-to-Moderate Acne. J Cosmet Dermatol. 2025 May;24(5):e70220. doi: 10.1111/jocd.70220. PMID 40321085